CLINICAL TRIAL: NCT03695497
Title: A Randomized Controlled Trial Comparing Direct Anterior Approach to Direct Lateral Approach in Patients Receiving a Total Hip Arthroplasty for Femoral Neck Fracture - a 1 Year Follow-up Study
Brief Title: Direct Anterior Approach for Femoral Neck Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Møre og Romsdal HF (Other Government)
Collaborators: St. Olavs Hospital (Other); Kristiansund Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/935
Record Dates: First submitted 2018-10-02; First posted 2018-10-04 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Femoral Neck Fractures
Keywords: Arthroplasty, Replacement, Hip; Orthopedic procedures
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Direct anterior approach (Experimental): total hip arthroplasty with direct anterior approach
  Interventions: Procedure: Direct anterior approach
- Direct Lateral Approach (Experimental): total hip arthroplasty with direct lateral approach
  Interventions: Procedure: Direct Lateral Approach

INTERVENTIONS:
Procedure: Direct anterior approach — total hip arthroplasty with DAA
  Other Names: DAA
  Arms: Direct anterior approach
Procedure: Direct Lateral Approach — total hip arthroplasty with DLA
  Other Names: DLA
  Arms: Direct Lateral Approach

SUMMARY:
The primary objective is to examine if in patients with a dislocated femoral neck fracture who receive a total hip arthroplasty, direct anterior approach will give a better result in terms of mobilization, function and pain in the first weeks and months postoperatively, than direct lateral approach.

DETAILED DESCRIPTION:
first included patient 23th November 2018

ELIGIBILITY:
Inclusion Criteria:

* Dislocated femoral neck fracture

Exclusion Criteria:

* Infection around the hip (soft tissue or bone)
* Pathologic fracture
* Excessive alcohol or substance abuse that most likely will give reduced compliance
* Patients with any fractures of the long bones in the lower extremity, fracture of the spine, and/or intra-thoracic or intra-abdominal injury (i.e., multiple trauma). Because the outcomes and clinical course of patients with multiple trauma may be quite different from a non-trauma patient.
* Bedridden patients/non-walkers
* Patients with an underlying illness that doesn't have life expectancy beyond six months
* In case of severe cognitive impairment where the patients are not able to give their informed consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Difference in Timed Up and Go Test (TUG) between the groups | 6 weeks postoperatively.
  It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.

SECONDARY OUTCOMES:
Difference in Forgotten Joint Score for hip (FJS-12) between the groups | 2,6,12 weeks, and 1 year
  12 questions. Every question is scored 1 (never) to 5 (mostly) according to the selected response categories. Thus, the raw score ranges from 12 to 60. The raw score is linearly transformed to a 0-100 scale and then reversed to obtain the final score. Final score = 100 - ((sum(item01 to item12) - 12)/48*100) For the final 'Forgotten Joint Score -12' a high score indicates good outcome.
Difference in EQ-5D-5L score between the groups | 2,6,12 weeks, and 1 year
  5 questions. Every question is scored 1 to 5 where 5 is worse outcome. For example one profile could be' 12233'. As there is no Norwegian index, the EQ5D-5L was converted into a Swedish index score.
Difference in Oxford Hip Score (OHS) between the groups | 2,6,12 weeks, and 1 year
  12 questions. Every question is scored 4 to 0 according to the selected response. Thus the highest score on 48 means a perfectly functioning hip, while a score on 0 means the worst outcome.
Difference in Timed Up and Go Test (TUG) between the groups | 2,12 weeks, 1 year.
  It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down
Difference in EQ5D-VAS between the groups | 2,6,12 weeks, and 1 year
  Respondents report their perceived health status with a grade ranging from 0 (worst possible health status) to 100 (best possible health status).
radiological results 1. | postoperative, 3,12 months.
  We will look at the offset of the hip prosthesis.
radiological results 2. | postoperative, 3,12 months.
  We will look at alignment of the stem. Femoral component angulation between 3° varus and 3° valgus relative to the femoral shaft axis will be considered neutral. Positioning outside this references will be graded as varus or valgus
radiological results 3. | postoperative, 3,12 months.
  We will look at quality of stem cementation by Barrack
radiological results 4. | postoperative, 3,12 months.
  We will look at leg length. It will be measured using the vertical height from the interteardrop line.
radiological results 5. | postoperative, 3,12 months.
  We will look at inclination of the cup.It will be measured in reference to the interteardrop line.
radiological results 6. | postoperative, 3,12 months.
  We will look at anteversion of the cup. It will be measured using the ischiolateral method.
complications | Within the first year postoperatively.
  periprosthetic fractures, dislocation, implant failure, neurovascular injury, infection. abductor failure, neurapraxia of LFCN), and mortality

OTHER OUTCOMES:
Change in CK (Creatine Kinase) | preoperatively and day 1,2,3,4 postoperatively.
  Measure CK preoperatively and the first 4 postoperative days.
Change in CRP (C-Reactive Protein) | preoperatively and day 1,2,3,4 postoperatively.
  Measure CRP preoperatively and the first 4 postoperative days.
Change in Hb (Hemoglobin)-levels. | preoperatively and day 1,2,3,4 postoperatively.
  Measure Hb preoperatively and the first 4 postoperative days.

CONTACTS AND LOCATIONS:
Overall Officials: Øystein B Lian, md phd, Study Chair — Helse Møre og Romsdal Hospital Trust (HF), Kristiansund Hospital
Locations (1):
- Kristiansund Hospital, Kristiansund, Norway

IPD SHARING:
Plan to Share IPD: No